## 

Study ID #: HSM#17-00775/IRB-17-01997 Form Version Date:10/23/2017

#### TITLE OF RESEARCH STUDY:

Title: EFFICACY OF TRANEXAMIC ACID IN FOOT AND ANKLE SURGERIES - A RANDOMIZED CONTROLLED TRIAL

### PRINCIPAL INVESTIGATOR (HEAD RESEARCHER) NAME AND CONTACT INFORMATION:

Name: Yan Lai, MD

Physical Address: Mount Sinai West, 1000 10th Avenue, New York, NY 10019

Mailing Address: Department of Anesthesiology Mount Sinai West 1000 10th Avenue, New York, NY

10019

Phone: 212-523-6915

#### WHAT IS A RESEARCH STUDY?

A research study is when scientists try to answer a question about something that we don't know enough about. Participating may not help you or others.

People volunteer to be in a research study. The decision about whether or not to take part is totally up to you. You can also agree to take part now and later change your mind. Whatever you decide is okay. It will not affect your ability to get medical care within the Mount Sinai Health System.

Someone will explain this research study to you. Feel free to ask all the questions you want before you decide. Any new information that develops during this research study that might make you change your mind about participating will be given to you promptly.

Basic information about this study will appear on the website http://www.ClinicalTrials.gov. There are a few reasons for this: the National Institutes of Health (NIH) encourages all researchers to post their research; some medical journals only accept articles if the research was posted on the website; and, for research studies the U.S. Food and Drug Administration (FDA) calls "applicable clinical trials" a description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

### PURPOSE OF THIS RESEARCH STUDY:

The purpose of our study is to evaluate if tranexamic acid, a medication which commonly helps promote blood clots if given intravenously reduces blood loss in patients undergoing foot and ankle.

This medication is routinely used in orthopedic surgeries to reduce blood loss during the surgery. Reduced blood loss avoids the need to blood transfusion and provides better operating conditions for the surgeon. Our study attempts to find out if tranexamic acid is effective in reducing blood loss in foot and ankle surgeries.

------FOR IRB USE ONLY-----------------------FOR IRB USE ONLY-------------------

### 

Study ID #: HSM#17-00775/IRB-17-01997

You may qualify to take part in this research study because you are a healthy individual between the ages of 18 and 75 undergoing foot and ankle surgery. Funds for conducting this research are

Form Version Date: 10/23/2017

# LENGTH OF TIME AND NUMBER OF PEOPLE EXPECTED TO PARTICIPATE

Your participation in this research study is expected to last from the day of surgery to first post operative visit at the surgeon's office.

The total number of people expected to take part in this research study is 200 participants.

#### **DESCRIPTION OF WHAT'S INVOLVED:**

provided by Mount Sinai.

If you agree to participate in this research study at the Mount Sinai West hospital, the following information describes what may be involved.

On the day of your surgery your anesthesia provider will perform a history and physical. This involves discussing your medical and surgical history and reviewing your allergies as well as your medications along with a focused physical exam. A small catheter, known as an intravenous (IV) line, will also be placed in one of your veins in preparation for your surgery.

After discussing the anesthetic plan with your anesthesia provider you will be entering the operating room. Based on which group you have been randomly assigned to, either tranexamic acid medication or placebo in the form of normal saline, will be administered to you by infusing through the intravenous catheter that was inserted in your vein(intravenous catheter or IV line),at the start of the procedure and towards the end of the procedure while you are under anesthesia. You will randomly be assigned to either of the treatment groups and each subject has an equal chance of being in either group. Randomization will occur via a computer software number generator that will assign you to either of the groups.

A placebo is a substance (in this case normal saline) with no therapeutic effect. You will randomly be assigned to either of the treatment groups and each subject has an equal chance of being in either group. If you have been assigned to the tranexamic acid group, you will have received tranexamic acid by intravenous method at the start of your surgery and towards the end while you are under anesthesia. If you have been assigned to the placebo group, you will receive a placebo (normal saline) at the start of your surgery and towards the end of the surgery while you are under anesthesia. All patients undergoing anesthesia are required to have an intravenous line placed. The amount of blood loss during your entire surgery will be recorded. Blood loss will be measured in terms of number of lap pads used and blood collected in the canister.

After surgery you will be transferred to the post anesthesia care unit (PACU) also known as the recovery room. Your pain scores will be assessed and treated.

The amount of blood loss during the first 24 hours during your hospital stay will be recorded. The number of days of hospitalization will be be recorded.

------FOR IRB USE ONLY------

## 

Form Version Date: 10/23/2017

Study ID #: HSM#17-00775/IRB-17-01997

During the first follow up visit at surgeon's office the following information like any associated wound complication, wound healing time, incidence of infection will be recorded. Your blood will be collected to assess blood counts also.

The use of tranexemic acid in orthopedic surgeries is currently the standard of care to reduce blood loss. There are currently no standards or guidelines for the preference of tranexamic acid in foot and ankle studies and its efficacy in reducing blood loss which is the focus of this research study.

The study treatment you get will be chosen by chance, like flipping a coin. Neither you nor the study doctor will choose what study treatment you get. You will have an equal chance of being given each study treatment. You will not be told which study treatment you are getting, however your study doctor will know.

#### YOUR RESPONSIBILITIES IF YOU TAKE PART IN THIS RESEARCH:

If you decide to take part in this research study you will be responsible for the following things: Your participation in this research study is expected to last from the time you meet your surgeon at his office, your anesthesia providers on the day of your surgery and until the first office visit back at your surgeon's office.

#### COSTS OR PAYMENTS THAT MAY RESULT FROM PARTICIPATION:

You will not be paid for participating in this research study. Being in this research study will not lead to extra costs to you. You will not be reimbursed for your travel or time that may be required for study visits.

#### **POSSIBLE BENEFITS:**

It is important to know that you may not get any benefit from taking part in this research. Others may not benefit either. However, possible benefits may be reduced blood loss during your surgery.

#### **REASONABLY FORESEEABLE RISKS AND DISCOMFORTS:**

Risk of loss of private information; this risk always exists, but there are procedures in place to minimize the risk.

As with any medication, there is a possibility of an allergic reaction. Although rare, possible complications include hypersensitivity reaction, bleeding or local site infection, thrombosis and chance of any vascular event. There is a possible risk of private information with procedures in place to minimize the risk.

#### OTHER POSSIBLE OPTIONS TO CONSIDER:

### 

Study ID #: HSM#17-00775/IRB-17-01997

You may decide not to take part in this research study without any penalty. The choice is totally up to

Form Version Date: 10/23/2017

you.

#### IN CASE OF INJURY DURING THIS RESEARCH STUDY:

If you believe that you have suffered an injury related to this research as a participant in this study, you should contact the Principal Investigator.

#### ENDING PARTICIPATION IN THE RESEARCH STUDY:

You may stop taking part in this research study at any time without any penalty. This will not affect your ability to receive medical care at any of the Mount Sinai Health System hospitals or to receive any benefits to which you are otherwise entitled.

If you decide to stop being in the research study, please contact the Principal Investigator or the research staff. You may also withdraw your permission for the use and disclosure of any of your protected information for research, but <u>you must do so in writing</u> to the Principal Investigator at the address on the first page. Even if you withdraw your permission, the Principal Investigator for the research study may still use the information that was already collected if that information is necessary to complete the research study. Your health information may still be used or shared after you withdraw your authorization if you have an adverse event (a bad effect) from participating in the research study.

<u>Withdrawal without your consent</u>: The study doctor, the sponsor or the institution may stop your involvement in this research study at any time without your consent. This may be because the research study is being stopped, the instructions of the study team have not been followed, the investigator believes it is in your best interest, or for any other reason. If specimens or data have been stored as part of the research study, they too can be destroyed without your consent.

#### **CONTACT PERSON(S):**

If you have any questions, concerns, or complaints at any time about this research, or you think the research has hurt you, please contact the office of the research team and/or the Principal Investigator at (212)-523-6915.

This research has been reviewed and approved by an Institutional Review Board. You may reach a representative of the Program for Protection of Human Subjects at the Icahn School of Medicine at Mount Sinai at telephone number (212) 824-8200 during standard work hours for any of the reasons listed below. This office will direct your call to the right person within the Mount Sinai Health System:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.

| FOR IRB USE ONLY |
|------------------|
|------------------|

### 

Form Version Date: 10/23/2017

Study ID #: HSM#17-00775/IRB-17-01997

- You are not comfortable talking to the research team.
- You have questions about your rights as a research subject.
- You want to get information or provide input about this research.

#### **DISCLOSURE OF FINANCIAL INTERESTS:**

Sometimes, physicians/researchers receive payments for consulting or similar work performed for industry. Effective September 2014 Mount Sinai reviews only payments to an individual totaling more than \$5,000 a year per entity when determining potential conflicts of interest. If you have questions regarding industry relationships, we encourage you to talk your physician/researcher or visit our website at http://icahn.mssm.edu/ where Mount Sinai publicly discloses the industry relationships of our faculty.

#### **MAINTAINING CONFIDENTIALITY - HIPAA AUTHORIZATION:**

As you take part in this research project it will be necessary for the research team and others to use and share some of your private protected health information. Consistent with the federal Health Insurance Portability and Accountability Act (HIPAA), we are asking your permission to receive, use and share that information.

What protected health information is collected and used in this study, and might also be disclosed (shared) with others?

As part of this research project, the research team at the hospital(s) involved in the research will collect your name, address, telephone number, and medical record number.

The researchers will also get information from your medical record including pertinent medical history, type of surgery and type of anesthesia delivered.

During the study the researchers will gather information by:

- taking a medical history (includes current and past medications or therapies, illnesses, conditions or symptoms, family medical history, allergies, etc.)
- doing a physical examination that generally also includes blood pressure reading, heart rate, breathing rate and temperature
- completing the tests, procedures, questionnaires and interviews explained in the description section of this consent.

#### Why is your protected health information being used?

Your personal contact information is important to be able to contact you during the study. Your health information and the results of any tests and procedures being collected as part of this research study will be used for the purpose of this study as explained earlier in this consent form. The results of this

-----FOR IRB USE ONLY-------

### 

Form Version Date: 10/23/2017

Study ID #: HSM#17-00775/IRB-17-01997

study could be published or presented at scientific meetings, lectures, or other events, but would not include any information that would let others know who you are, unless you give separate permission to do so.

The Principal Investigator may also use and share the results of these tests and procedures to treat you in collaboration with others in the Mount Sinai Health System.

The research team and other authorized members of The Mount Sinai Health System ("Mount Sinai") workforce may use and share your information to ensure that the research meets legal, institutional or accreditation requirements. For example, the School's Program for the Protection of Human Subjects is responsible for overseeing research on human subjects, and may need to see your information. If you receive any payments for taking part in this study, the Mount Sinai Finance Department may need your name, address, social security number, payment amount, and related information for tax reporting purposes. If the research team uncovers abuse, neglect, or reportable diseases, this information may be disclosed to appropriate authorities.

#### Who, outside Mount Sinai, might receive your protected health information?

As part of the study, the Principal Investigator, study team and others in the Mount Sinai workforce may disclose your protected health information, including the results of the research study tests and procedures, to the following people or organizations: (It is possible that there may be changes to the list during this research study; you may request an up-to-date list at any time by contacting the Principal Investigator.)

- Other collaborating research center(s) and their associated research/clinical staff who are working with the investigators on this project: Mount Sinai Hospital, Mount Sinai St. Luke's
- A Data Safety Monitoring Board or other committee that will monitor the study on an ongoing basis for safety.
- The United States Department of Health and Human Services and the Office of Human Research Protection.

In all disclosures outside of Mount Sinai, you will not be identified by name, social security number, address, telephone numbers or any other direct personal identifier unless disclosure of the direct identifier is required by law. Some records and information disclosed may be identified with a unique code number. The Principal Investigator will ensure that the key to the code will be kept in a locked file, or will be securely stored electronically. The code will not be used to link the information back to you without your permission, unless the law requires it, or rarely if the Institutional Review Board allows it after determining that there would be minimal risk to your privacy. It is possible that a sponsor or their representatives, a data coordinating office, a contract research organization, may come to inspect your records. Even if those records are identifiable when inspected, the information leaving the institution will be stripped of direct identifiers. Additionally, when applicable, the monitors, auditors, the IRB, the Office of Human Subjects Protection (OHRP) of the Department of Health and Human Services as well as the Food and Drug Administration (FDA) will be granted direct access to

### 

Form Version Date: 10/23/2017

Study ID #: HSM#17-00775/IRB-17-01997

your medical records for verification of the research procedures and data. OHRP and FDA are authorized to remove information with identifiers if necessary to complete their task. By signing this document you are authorizing this access. We may publish the results of this research. However, we will keep your name and other identifying information confidential.

For how long will Mount Sinai be able to use or disclose your protected health information? Your authorization for use of your protected health information for this specific study does not expire.

#### Will you be able to access your records?

During your participation in this study, you will not be able to access your medical records. This will be done to prevent the knowledge of study results from affecting the reliability of the study. Your information will be available should an emergency arise that would require your treating physician to know this information to best treat you. You will have access to your medical record and any study information that is part of that record when the study is over or earlier, if possible. The investigator is not required to release to you research information that is not part of your medical record.

#### Do you need to give us permission to obtain, use or share your health information?

NO! If you decide not to let us obtain, use or share your health information you should not sign this form, and you will not be allowed to volunteer in the research study. If you do not sign, it will not affect your treatment, payment or enrollment in any health plans or affect your eligibility for benefits.

### Can you change your mind?

You may withdraw your permission for the use and disclosure of any of your protected information for research, but you must do so in writing to the Principal Investigator at the address on the first page. Even if you withdraw your permission, the Principal Investigator for the research study may still use your protected information that was already collected if that information is necessary to complete the study. Your health information may still be used or shared after you withdraw your authorization if you should have an adverse event (a bad effect) from being in the study. If you withdraw your permission to use your protected health information for research that means you will also be withdrawn from the research study, but standard medical care and any other benefits to which you are entitled will not be affected. You can also tell us you want to withdraw from the research study at any time without canceling the Authorization to use your data.

If you have not already received it, you will also be given The Hospital's Notice of Privacy Practices that contains more information about how The Hospital uses and discloses your protected health information.

It is important for you to understand that once information is disclosed to others outside Mount Sinai, the information may be re-disclosed and will no longer be covered by the federal privacy protection regulations. However, even if your information will no longer be protected by federal regulations, where possible, Mount Sinai has entered into agreements with those who will receive your information to continue to protect your confidentiality.

If as part of this research project your medical records are being reviewed, or a medical history is being taken, it is possible that HIV-related information may be revealed to the researchers. If that is

## 

Study ID #: HSM#17-00775/IRB-17-01997

be ignored.

the case, the following information concerns you. If this research does not involve any review of medical records or questions about your medical history or conditions, then the following section may

Form Version Date: 10/23/2017

## **Notice Concerning HIV-Related Information**

If you are authorizing the release of HIV-related information, you should be aware that the recipient(s) is (are) prohibited from re-disclosing any HIV-related information without your authorization unless permitted to do so under federal or state law. You also have a right to request a list of people who may receive or use your HIV-related information without authorization. If you experience discrimination because of the release or disclosure of HIV-related information, you may contact the New York State Division of Human Rights at (888) 392-3644 or the New York City Commission on Human Rights at (212) 306-5070. These agencies are responsible for protecting your rights.


Study ID #: HSM#17-00775/IRB-17-01997 Form Version Date:10/23/2017

| Your signature below documents your permission to take part in the disclosure of your protected health information. A signed and dated | |
|---|---|
| Signature of subject | Date |
| Printed name of subject | Time |
| Person Explaining Study and Obtaining 0 | Consent |
| Signature of person obtaining consent | Date |
| Printed name of person obtaining consent | Time |
| Witness Section: For use when a witness is required to or document below (for example, subject is illiterate or visually in short form consent): My signature below documents that the information in the consent written information was accurately explained to, and apparently unotated that consent was freely given by the subject. | npaired, or this accompanion document and any other |
| Signature of witness to consent process | Date |
| Printed name of person witnessing consent process | Time |
| FOR IRB USE ONLY | |

Rev6.22.16